CLINICAL TRIAL: NCT04443400
Title: Early Detection of Cardiac Damage by Two-Dimensional Speckle Tracking Echocardiography After Thoracic Radiation Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUTN
Record Dates: First submitted 2020-06-21; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Radiation Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — blood samples will be collected
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to detecte and predict early subclinical cardiac damage induced by thoracic radiation therapy based on two-dimensional speckle tracking echocardiography combined with multiple circulating biomarkers.

DETAILED DESCRIPTION:
This is a monocentric prospective cohort study in which 100 patients treated for malignant tumors and with cardiac radiation exposure will be included.All patient will be followed for 12 months after radiotherapy. Echocardiography, 2D STE parameters and circulating biomarkers will be collected.

ELIGIBILITY:
Inclusion Criteria:

* with malignant tumors
* will receive radiotherapy
* with cardiac exposure during the radiotherapy process
* could receive regular follow-up for 12 months
* written informed consent

Exclusion Criteria:

* satisfactory echocardiographic images could not be obtained
* moderate or severe valvular disease
* cardiomyopathy
* congenital heart disease
* refractory hypertension
* coronary artery disease*
* heart failure
* arrhythmia requiring intervention
* pericarditis
* acute myocarditis
* participating in other clinical studies of drug intervention
* severe liver and kidney dysfunction
* autoimmune disease
* pulmonary hypertension

coronary artery disease: at least 50% stenosis besed on previous coronary angiography or CTA, or with a history of percutaneous coronary stent implantation.

*: with LVEF<50%, unstable angina，or acute myocardial infarction within 3 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with thoracic radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Early Detection of Cardiac Damage by Two-Dimensional Speckle Tracking Echocardiography After Thoracic Radiation Therapy | 2020-2021
  To detecte early subclinical cardiac damage induced by thoracic radiation therapy, based on two-dimensional speckle tracking echocardiography combined with multiple circulating biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Dan Zhu, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li T, Zhuang H, Wang Y, Li J, Zhu D, Cui M. Two-dimensional speckle tracking echocardiography in evaluating radiation-induced heart damage. Asia Pac J Oncol Nurs. 2021 Dec 25;9(2):119-124. doi: 10.1016/j.apjon.2021.12.008. eCollection 2022 Feb. PMID 35529415
- [Derived] Zhu D, Li T, Zhuang H, Cui M. Early Detection of Cardiac Damage by Two-Dimensional Speckle Tracking Echocardiography After Thoracic Radiation Therapy: Study Protocol for a Prospective Cohort Study. Front Cardiovasc Med. 2022 Jan 26;8:735265. doi: 10.3389/fcvm.2021.735265. eCollection 2021. PMID 35155592